CLINICAL TRIAL: NCT06032897
Title: The Effect of Personalized Music on the Elderly With Cognitive Impairment and Dementia: a Quasi-experimental Study.
Brief Title: Impact of Individualized Music Listening for People With Dementia on Anxiety: A Quasi-experimental Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: KMUHIRB-SV(Ⅰ)-20220050
Record Dates: First submitted 2023-08-28; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Music Listening
Keywords: dementia; individualized music listening; anxiety; behavior
MeSH Terms: conditions — Dementia; Anxiety Disorders; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): The control group who participated in routine activities
- experimental group (Experimental): The earphones were placed on individuals in the experimental group to listen to individualized music for 20 minutes. The individualized music listening were performed twice a week for four weeks, for a total of eight times.
  Interventions: Other: Individualized music listening (IML)

INTERVENTIONS:
Other: Individualized music listening (IML) — The earphones were placed on individuals in the experimental group to listen to individualized music for 20 minutes. The Individualized music listening (IML) were performed twice a week for four weeks, for a total of eight times.
  Arms: experimental group

SUMMARY:
This pilot study was designed to evaluate the effects of Individualized music listening (IML) implemented on older adults with mild cognitive impairment (MCI) and PwD. This quasi-experimental study used convenience sampling where thirty-two elderly individuals were recruited from five community-based dementia care centers then assigned to experimental (EG, n = 16) or control (CG, n = 16) groups according to the self-reports of importance of music in their lives and according to their personal wishes. The EG received eight treatments of IML (two times per week, 20 minutes per time), while the CG received the usual activities of the care centers for four weeks when EG received IML. The anxiety levels of both groups were investigated before and after first time IML and after eighth time IML. The researcher observed positive and negative behaviors of EG before, during and after each IML per 20 minutes in each time IML.

ELIGIBILITY:
Inclusion Criteria:

1. 50 years or older;
2. Mild cognitive impairment or dementia.

Exclusion Criteria:

1. Can not answer questions by themselves;
2. Have the habit of listening music in the past week.

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-08-25 (Actual); Primary Completion 2023-01-05 (Actual); Study Completion 2023-07-03 (Actual)

PRIMARY OUTCOMES:
Anxiety | First day: before the first time individualized music listening; first day: after completing first-time individualized music listeningof 20 minutes; the fourth week: after the last (eighth) time Individualized music listening of 20 minutes.
  The Chinese Mandarin version State-Trait Anxiety Inventory Y form. The scores of the 20 questions are summed with total score ranging from 20 to 80 points. The higher the total score, the higher the anxiety level.
Behavioral | Four weeks: eight times of individualized music listening. Before 20 minutes, during 20 minute, after 20 minute of every time individualized music listening.
  The Behavioral Observation Form for Intervention Condition checklist. If the 15 behaviors occurred in each period (20 minutes), the behavior column will be counted as 1 point in this time period, and if there were no behavior, it would be scored as 0 points. In this study, 15 behaviors were further classified into positive and negative behaviors (four negative behaviors included eye movement, agitation/restlessness, alertness, and sleeping), and then the scores of the two types of behaviors were summed up and the total score represented the performances of the behavior type. Higher scores mean more the type.

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Chao Lin, Principal Investigator — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University, Kaohsiung City, Taiwan